CLINICAL TRIAL: NCT00855348
Title: PRESEPT Study: Prospective Evaluation of Septin 9 Performance for Colorectal Cancer Screening
Brief Title: PRESEPT Study: Evaluation of SEPT9 Biomarker Performance for Colorectal Cancer Screening
Acronym: PRESEPT
Status: Completed | Type: Observational
Sponsor: Epigenomics, Inc (Industry)
Responsible Party: Timothy R. Church, Ph.D., University of Minnesota School of Public Health
Other Study IDs: Epigenomics_SPR0006
Record Dates: First submitted 2009-02-04; First posted 2009-03-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; early detection; methylation, biomarker
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Biomarkers; Blood Specimen Collection; DNA Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Eligible consented Subjects meeting inclusion / exclusion criteria will have 40 ml of blood drawn prior to undergoing bowel cleansing in preparation for screening colonoscopy. Subject blood specimens will be processed according to Epigenomics' plasma preparation procedure (Blood Collection and Plasma Preparation SOP.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults > 50 Years Scheduled for Colonscopy: Average to increased risk adults older than 50 years without symptoms indicative of CRC and designated for colonoscopy.
  Interventions: Other: All eligible subjects will provide blood for SEPT9 biomarker testing

INTERVENTIONS:
Other: All eligible subjects will provide blood for SEPT9 biomarker testing — A single blood sample per participant selected according to analysis plan is tested for evidence of methylation of a specific DNA sequence, SEPT9.
  Other Names: biomarker; blood; colorectal cancer; DNA methylation

SUMMARY:
The purpose of this study is to collect blood specimens and clinical data from screening guideline eligible individuals designated by their physician to receive a screening colonoscopy, and to evaluate the performance of a colorectal cancer-specific DNA methylation biomarker for detection of colorectal cancer in this cohort. Based on the outcome of the colonoscopy, polypectomy, biopsy and surgical tissue histopathology, the clinical utility of Septin 9 as colorectal cancer screening test will be evaluated.

DETAILED DESCRIPTION:
The study is designed as a prospective, open enrollment clinical investigation involving multiple clinical study sites in the United States and Germany. Subjects will be competitively enrolled at multiple sites until at least 50 invasive colorectal adenocarcinoma cases identified by screening colonoscopy and verified by clinical and histopathological examination have been enrolled. The primary objective of the investigation is to evaluate and describe the clinical performance of the Septin 9 Biomarker for detecting the 50 individuals with invasive colorectal adenocarcinoma identified in this population representative of the US screening guideline eligible population. Secondary objectives will be to evaluate and describe performance characteristics of the biomarker in individuals with adenomatous polyps 10 mm or larger, flat lesion (s) or non-invasive adenocarcinoma.

Collaborating sites will identify and contact patients scheduled for screening colonoscopy. These patients may be screened by the PI or designee to determine the patients' appropriateness for, and interest in, study participation. Study site personnel will meet with patients meeting eligibility guidelines and offer them participation. Patients interested in participation and who provide written informed consent will be enrolled as Subjects in the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent provided
* Capable of providing adequate health history
* Age 50 or older at time of colonoscopy (colorectal screening guideline eligible)
* Accessible for blood draw prior to start of bowel preparation for colonoscopy
* First large bowel endoscopy in lifetime

Exclusion Criteria:

* Anorectal bleeding or hematochezia within last 6 months for which patient sought medical attention
* Known iron deficiency anemia in the last 6 months for which patient sought medical attention
* Previous history of colorectal polyps or CRC
* High risk for colorectal cancer (2 or more 10 relatives with CRC; 1 or more 10 relative(s) < 50 years with CRC; known HNPCC or FAP)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in Subjects scheduled for screening colonoscopy according to current U.S. CRC screening guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 7929 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Clinical/surgical diagnosis of invasive colorectal adenocarcinoma detected by optical colonoscopy and confirmed by histology compared to the Septin 9 Biomarker classification. | One Year

SECONDARY OUTCOMES:
Detection of adenomatous polyp(s) equal to or greater than 10 mm, flat lesion (s) or non-invasive adenocarcinoma by colonoscopy and confirmed by histology compared to the Septin 9 Biomarker classification will also be described. | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Timothy R Church, Ph.D., Principal Investigator — University of Minnesota; Michael Wandell, PharmD., Study Director — Epigenomics, Inc; David F Ransohoff, MD, Study Chair — University of North Carolina
Locations (23):
- United States (20):
  - Digestive Care, Boca Raton, Florida
  - GI Care Center, Miami, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - Heartland Medical Research, Inc., Clive, Iowa
  - University of Louisville, Louisville, Kentucky
  - Minnesota Gastroenterology, Minneapolis, Minnesota
  - Jackson Gastrointestinal Associates, Jackson, Mississippi
  - Asheville Gastroenterology Associates PA, Asheville, North Carolina
  - Southern Gastroenterology Associates, New Bern, North Carolina
  - Digestive Health Specialists, Winston-Salem, North Carolina
  - The Portland Clinic, Portland, Oregon
  - Northwest Gastroenterology Clinic, Portland, Oregon
  - The Oregon Clinic, Portland, Oregon
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Medical University of South Carolina Digestive Disease Center, Charleston, South Carolina
  - Gastroenterology Center of the MidSouth, Germantown, Tennessee
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - Tacoma Digestive Disease Research Center, Tacoma, Washington
- Germany (3):
  - Berlin Private-Practice Gastroenterology Working Group, Berlin
  - University of Hamburg-Eppendorf, Hamburg
  - Technical University of Munich, Munich

REFERENCES:
- [Derived] Payne SR, Church TR, Wandell M, Rosch T, Osborn N, Snover D, Day RW, Ransohoff DF, Rex DK. Endoscopic detection of proximal serrated lesions and pathologic identification of sessile serrated adenomas/polyps vary on the basis of center. Clin Gastroenterol Hepatol. 2014 Jul;12(7):1119-26. doi: 10.1016/j.cgh.2013.11.034. Epub 2013 Dec 10. PMID 24333512
- [Derived] Church TR, Wandell M, Lofton-Day C, Mongin SJ, Burger M, Payne SR, Castanos-Velez E, Blumenstein BA, Rosch T, Osborn N, Snover D, Day RW, Ransohoff DF; PRESEPT Clinical Study Steering Committee, Investigators and Study Team. Prospective evaluation of methylated SEPT9 in plasma for detection of asymptomatic colorectal cancer. Gut. 2014 Feb;63(2):317-25. doi: 10.1136/gutjnl-2012-304149. Epub 2013 Feb 13. PMID 23408352